CLINICAL TRIAL: NCT04397341
Title: A Phase II Study of Biweekly Induction Regimen With Docetaxel, Cisplatin and Fluorouracil for Patients With Locally Advanced Squamous Cell Carcinoma of Head and Neck
Brief Title: Biweekly TPF Induction Chemotherapy for Locally Advanced Squamous Cell Carcinoma of Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Ching Yun Hsieh, Division of Hematology and Oncology, Department of internal medicine, China Medical University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH-HO-NPC001
Record Dates: First submitted 2020-05-17; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Locally Advanced Head and Neck Carcinoma
MeSH Terms: interventions — Docetaxel; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- biweekly TPF induction (Experimental): Docetaxel: 50 mg/m2 Cisplatin : 50 mg/m2 5-fluorouracil : 2,500 mg/m2 for 40-48 hrs Leucovorin: 250 mg/m2
  Interventions: Drug: docetaxel, cisplatin, fluorouracil

INTERVENTIONS:
Drug: docetaxel, cisplatin, fluorouracil — Biweekly Induction regimen with Docetaxel, Cisplatin and Fluorouracil

SUMMARY:
This study aimed to assess the efficacy and safety for biweekly TPF as induction chemotherapy for locally advanced head and neck cancer

DETAILED DESCRIPTION:
After being informed the study and potential risk, patients was provided written informed consent prior to initiating therapy. The chemotherapy regimen including docetaxel, cisplatin, 5-fluorouracil, and leucovorin was administered every 14 days for six cycles or until disease progression or intolerant treatment toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has histopathologically or cytologically confirmed diagnosis of stage 3 or 4 squamous cell carcinoma of the oral cavity, larynx, oropharynx or hypopharynx.
2. The patient has local advanced, and no distant metastatic, and unresectable disease.
3. The patient has measurable or valuable disease. 4 Age ≥ 20 years.

5. ECOG performance status 0, 1 or 2 at study entry. 6. Life expectancy ≥ 3 months. 7. The patient must have adequate organ function, defined as: 7a Absolute neutrophil count (ANC) ≥ 1.5 x 109/L; Platelets ≥ 100 x 109/L; Hemoglobin

* 9.0 g/dL. 7b Total Bilirubin ≤ 1.5 times upper limit of normal (ULN); Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN. 7c Alkaline phosphatase ≤ 2.5 x ULN. 7d Serum creatinine ≤ 1 x ULN or creatinine clearance ≥ 60 mL/min/1.73 m2. 8. Signed informed consent. 9 Women of child-bearing potential and men must be willing and able practice adequate contraception prior to study entry and for the duration of study treatment.

Exclusion Criteria:

1. The patient had previous chemotherapy or radiotherapy for squamous cell carcinoma of head and neck.
2. The patient has uncontrolled disorder(s), serious illness or medical condition(s) is/are not be enrolled to study that be confirmed by investigator.
3. Previous or concurrent malignancy except for basal or squamous cell skin cancer and/or in situ carcinoma of the cervix, or other solid tumors treated and without evidence of recurrence for at least 3 years prior to the study.
4. Peripheral neuropathy > Grade 2.
5. The patient is pregnant or breastfeeding.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2016-08-30 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Response rate after induction chemotherapy | through study completion, an average of 1 years
  CT and PET scan according to the RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Progression survival | Through study completion, an average of 6 months
  The time from the study registration date to the first day of disease progression at any site
Overall survival | Through study completion, an average of 6 months
  The time from the study registration date to the day of the patients' death.
Adverse event | through study completion, an average of 6 months
  Record adverse event

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsieh CY, Lein MY, Yang SN, Wang YC, Lin YJ, Lin CY, Hua CH, Tsai MH, Lin CC. Dose-dense TPF induction chemotherapy for locally advanced head and neck cancer: a phase II study. BMC Cancer. 2020 Sep 1;20(1):832. doi: 10.1186/s12885-020-07347-6. PMID 32873270